CLINICAL TRIAL: NCT02454699
Title: A Phase 1 Trial to Evaluate the Safety and Pharmacokinetics of Multiple Ascending Doses of MBX-400 in Healthy Volunteers
Brief Title: Safety and PK of MBX-400 (Cyclopropavir) in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0092; HHSN272201300018I
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-07-19

CONDITIONS: Cytomegalovirus Infection
Keywords: antiviral; ascending dose; Cytomegalovirus; food effect; Herpesviridae; MBX-400
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1000mg MBX400 (Experimental): 6 subjects receive 1000 mg MBX400 orally once per day for 7 days, 2 subjects receive Placebo orally once per day for 7 days
  Interventions: Drug: MBX400; Other: Placebo
- 100mg MBX400 (Experimental): 6 subjects receive 100 mg MBX400 orally once per day for 7 days, 2 subjects receive Placebo orally once per day for 7 days
  Interventions: Drug: MBX400; Other: Placebo
- 350mg MBX400 (Experimental): 6 subjects receive 350 mg MBX400 orally once per day for 7 days, 2 subjects receive Placebo orally once per day for 7 days
  Interventions: Drug: MBX400; Other: Placebo
- 750mg MBX400 (Experimental): 6 subjects receive 750 mg MBX400 orally once per day for 7 days, 2 subjects receive Placebo orally once per day for 7 days
  Interventions: Drug: MBX400; Other: Placebo

INTERVENTIONS:
Drug: MBX400 — MBX-400, a white to off-white crystalline powder, will be given orally x 7 days to 4 cohorts. Cohort 1 receives 100 mg/day, Cohort 2 receives 350 mg, Cohort 3 receives 750 mg, Cohort 4 receives 1000 mg.
Other: Placebo — Placebo capsules are supplied as white opaque, hard gelatin capsules filled with microcrystalline cellulose. 2 subjects from each cohort receive Placebo orally once per day x 7 days.

SUMMARY:
This is a phase I safety, PK and food effect study of the CMV drug. In part 1 of the study, subjects will receive one of four dosage strengths of MBX-400 (100 mg once daily, 350 mg once daily; 750 mg once daily; and 1000 once daily) for 7 days and safety and PK will be assessed. Subjects must be 18 to 65 years of age, male or female; if female, be surgically-sterilized or post-menopausal; if male, have undergone vasectomy; have a body mass index (BMI) of 18 to 32 kg/m^2; not be a user of nicotine-containing products; be willing to abstain from nicotine-containing products, alcohol and illicit drugs during the study. Subjects will be followed for 28 days post dosing.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a common cause of viral illness in children and adults. CMV is also an important congenital infection with complications including deafness, developmental delay, and cerebral palsy. The proposed study design is a standard multiple ascending dose escalation study. Four cohorts of 8 subjects each (6 active; 2 placebo) will be enrolled sequentially. MBX-400 will be administered orally once daily for 7 days, in the form of capsules, by study staff while the subject is an inpatient in a research unit. The study doses will be 100, 350, 750, and 1,000 mg daily. Up to 32 healthy male and female (non-pregnant, non-lactating) volunteers ages 18-65 in one site, will be consented and allowed to participate in the study if upon screening they meet the inclusion/exclusion criteria. Subjects will be enrolled into one of four sequential cohorts groups: Cohort 1 will receive 100 mg PO once daily for 7 days, Cohort 2 will receive 350 mg PO once daily for 7 days, Cohort 3 will receive 750 mg PO once daily for 7 days, and Cohort 4 will receive 1000 mg PO once daily for 7 days of MBX-400. Two members of each cohort will receive placebo. The study duration for each subject is expected to be approximately 80 days (screening period, administration of daily dose, and follow-up). Each subject may be admitted to the unit 1 day prior to the first dose, and will remain in the unit until the day after the 7th daily dose. Subjects will return for follow-up visits after the last dose. Safety, tolerability, and pharmacokinetics will be assessed. The overall study duration across all study groups is expected to be approximately 18 months. The primary objective evaluate the safety and tolerability of multiple ascending doses of 100, 350, 750, and 1000 mg PO once daily for 7 days of MBX-400 in healthy subjects. The secondary objective determine the plasma and urine pharmacokinetic profile of multiple doses of 100, 350, 750, and 1000 mg PO once daily for 7 days of MBX-400 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide informed consent; 2. Subject age is between 18 through 65 years of age, inclusive; 3. Good general health as judged by the investigator; 4. Body Mass Index (BMI) between 18 to 32 kg/m^2; 5. Males or females who have either no capability or no sexual behavior that could result in fathering or conceiving a child in the future; Meeting this inclusion criterion would be demonstrated by one of the parameters below: -Surgical sterilization (vasectomy, tubal ligation, or hysterectomy) -Females who are post-menopausal, as defined by the absence of menstrual periods for greater than one year after age 45 without alternate diagnosis (e.g., PCOS) -Absence of any heterosexual activity except with a partner meeting one of the above criteria; 6. Available and willing to participate in the study procedures and requirements; Able and willing to stay in a clinical facility for up to 10 days and return for all visits; swallow the capsules provided; and have blood and urine collections for the duration of the study. 7. Non-smoker, former smoker, or former user of nicotine-containing products Former smoker/user defined as someone who smoked or used nicotine-products one or more times a week for at least one month who has not smoked for at least 3 months and has not used nicotine-containing products for at least 1 month and is willing to abstain from nicotine-containing products during the study; 8. Willing to abstain from alcohol until after Day 10 visit* and should moderate drinking through study end (less than or equal to 2 drinks/day). Illicit drugs should not be used throughout the study; *the completion of PK collections 9. Demonstrates knowledge and comprehension of the study by passing a questionnaire of the study protocol with a score of at least 70%. Anyone not passing the test initially may retake the test once.

Exclusion Criteria:

1.Have had an acute illness and/or an oral temperature >100.4°F (38°C) within three days prior to drug dosing; 2.Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation; Including acute or chronic medical disease or condition, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study. 3.Have a known allergy to the components of MBX-400 or placebo capsules (microcrystalline cellulose, gelatin, titanium dioxide); 4.Have a history of anaphylaxis or other serious adverse reactions to nucleoside analog medications; 5.Have an active malignancy or history of metastatic or hematologic malignancy; 6.Have clinically significant abnormal ECG at screening based on ECG reading by pre-defined study consulting cardiologist; Including: 1) conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS> / =120ms, PR> / =220ms, any second or third degree AV block, or QTc prolongation (>450ms); 2) significant repolarization (ST segment or T wave) abnormality; 3) significant atrial or ventricular arrhythmia; 4) frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, 2 premature ventricular contractions in a row); 5) ST elevation consistent with ischemia; or 6) evidence of past or evolving myocardial infarction 7.Have known currently active HIV, CMV, hepatitis B or hepatitis C infection; 8.Have clinically significant anemia or bleeding disorder; 9.Have clinically significant gastrointestinal disorder including ulcer disease or conditions affecting absorption; 10.Have a blood pressure or heart rate that is a Grade > / =1; 11.Have a total White Blood Cell (WBC) count, Absolute Neutrophil Count (ANC), hemoglobin or platelet count that is a Grade > / =1 at screening; 12.Have a creatinine higher than the normal range at screening; 13.Have an Alanine Aminotransferase (ALT) or an Aspartate Aminotransferase (AST) > Upper Limit of Normal at screening; 14.Have PT or PTT that is a Grade > / =1 at screening; 15.Have any electrolyte level (sodium, potassium) that is a Grade > / =1 at screening; 16.Have a value higher than trace for glucose, hemoglobin and/or protein on urinalysis at screening; 17.Have ongoing drug abuse/dependence (including alcohol) or a history of this within five years of enrollment; 18.Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other major psychiatric diagnosis; 19.Have a history of hospitalization for psychiatric illness, suicide attempt, or confinement for danger to self or others, within the past 10 years; Subjects with a psychiatric disorder not meeting exclusion criteria, e.g., attention-deficit hyperactivity disorder, that is controlled for a minimum of 3 months may be enrolled as long as the investigator has determined that the subject's mental status will not compromise the subject's ability to comply with protocol. 20.Have donated blood within 30 days prior to Day 1 or plans to donate blood during the study; 21.Have taken any drug active against herpes viruses within 30 days prior to Day 1 including but not limited to: acyclovir, valacyclovir, famciclovir, penciclovir, ganciclovir and valganciclovir; 22.Use of any medication on a chronic basis; 23.Use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages within 72 hours prior to Check-in (Day -1); 24. Are taking or have utilized any drugs within 3 days prior to Day 1; alcohol or tobacco within 3 days prior to Day 1; or are a chronic alcohol user; Concomitant medications, including prescription and over the counter medications as well as herbals, vitamins and supplements, are not allowed within 3 days prior to Day 1. Chronic alcohol user is defined as consuming 10 or more alcoholic drinks per week. 25.Urine cotinine level >150 ng/mL; 26.Have taken any investigational agents within 28 days of Day 1; 27.Have a positive urine drug screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Frequency of clinical and laboratory adverse events and serious adverse events related to the study product through Day 22. | Day 1 through Day 22

SECONDARY OUTCOMES:
Amount of drug excreted in urine with dose 1 | Day 1 pre-dose, 0-4, 4-8, 8-12, and 12-24 hour collections
Amount of drug excreted in urine with dose 7 | Day 7 pre-dose, 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72 hour collections
Drug accumulation ratio | Between Days 1 and 7
Pharmacokinetic characteristics of MBX-400: amount excreted in urine (Ae) | Day 1 dose at baseline pre-dose and the following intervals: 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours. Day 7 dose: baseline pre-dose and the following intervals: 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-48 hours, and 48-72 hours.
Pharmacokinetic characteristics of MBX-400: AUC0-inf | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing
Pharmacokinetic characteristics of MBX-400: CI/F | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing
Pharmacokinetic characteristics of MBX-400: Cmax | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing
Pharmacokinetic characteristics of MBX-400: drug accumulation ratio between days 1 and 7. | Days 1 through 7
Pharmacokinetic characteristics of MBX-400: t1/2 | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing
Pharmacokinetic characteristics of MBX-400: Tmax | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing
Pharmacokinetic characteristics of MBX-400: total urine collection and clearance (Clu) | Day 1 dose at baseline pre-dose and the following intervals: 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours. Day 7 dose: baseline pre-dose and the following intervals: 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-48 hours, and 48-72 hours.
Pharmacokinetic characteristics of MBX-400: Vd/F | 8 time-points over 24 hours after dosing on Day 1; immediately pre-dose and 2 hours after dosing on day 4; and on day 7 at 8 time-points over 24 hours, then at 30, 48, and 72 hours after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Vaccine Center - The Hope Clinic, Decatur, Georgia, United States

REFERENCES:
- [Derived] Rouphael NG, Hurwitz SJ, Hart M, Beck A, Anderson EJ, Deye G, Osborn B, Cai SY, Focht C, Amegashie C, Bowlin TL, Brooks J, Mulligan MJ. Phase Ib Trial To Evaluate the Safety and Pharmacokinetics of Multiple Ascending Doses of Filociclovir (MBX-400, Cyclopropavir) in Healthy Volunteers. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00717-19. doi: 10.1128/AAC.00717-19. Print 2019 Sep. PMID 31285228